CLINICAL TRIAL: NCT01547598
Title: Safety and Efficacy of LUMIGAN® RC Versus DuoTrav® in Patients Who Require Further Intraocular Pressure (IOP) Reduction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMA-LUM-11-020
Record Dates: First submitted 2012-02-10; First posted 2012-03-08 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost; Timolol; Duotrav

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LUMIGAN® RC (Active Comparator): Travatan® Z (travoprost ophthalmic solution 0.004%) administered as 1 drop in the affected eye(s) once a day for 4 weeks. Then, LUMIGAN® RC (bimatoprost ophthalmic solution 0.01%) administered as 1 drop in the affected eye(s) once daily in the evening for 12 weeks.
  Interventions: Drug: travoprost ophthalmic solution 0.004%; Drug: Bimatoprost ophthalmic solution 0.01%
- DuoTrav® (Active Comparator): Travatan® Z (travoprost ophthalmic solution 0.004%) administered as 1 drop in the affected eye(s) once a day for 4 weeks. Then, DuoTrav® (travoprost 0.004% / timolol 0.5% combination ophthalmic solution) administered as 1 drop in the affected eye(s) once daily in the morning for 12 weeks.
  Interventions: Drug: travoprost ophthalmic solution 0.004%; Drug: travoprost 0.004% / timolol 0.5% combination ophthalmic solution

INTERVENTIONS:
Drug: travoprost ophthalmic solution 0.004% — Travatan® Z (travoprost ophthalmic solution 0.004%) administered as 1 drop in the affected eye(s) once a day for 4 weeks.
  Other Names: Travatan® Z
Drug: travoprost 0.004% / timolol 0.5% combination ophthalmic solution — DuoTrav® (travoprost 0.004% / timolol 0.5% combination ophthalmic solution) administered as 1 drop in the affected eye(s) once daily in the morning for 12 weeks.
  Other Names: DuoTrav®
  Arms: DuoTrav®
Drug: Bimatoprost ophthalmic solution 0.01% — LUMIGAN® RC (bimatoprost ophthalmic solution 0.01%) administered as 1 drop in the affected eye(s) once daily in the evening for 12 weeks.
  Other Names: LUMIGAN® RC
  Arms: LUMIGAN® RC

SUMMARY:
This non-inferiority study will assess safety and efficacy of LUMIGAN® RC (bimatoprost ophthalmic solution 0.01%) versus DuoTrav® (travoprost 0.004%/timolol 0.5% combination ophthalmic solution) in patients previously on Travatan® Z (travoprost ophthalmic solution 0.004%) monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Open angle glaucoma or ocular hypertension
* Best corrected visual acuity of 20/100 or better in both eyes

Exclusion Criteria:

* Ocular surgery within 3 months, or anticipated ocular surgery within 12 weeks
* Previous treatment with LUMIGAN® RC or DuoTrav®
* History of LASIK, LASEK, RK or PRK in the study eye(s)
* Active ocular inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LUMIGAN® RC | DuoTrav®
Started | 67 | 68
Completed | 61 | 63
Not Completed | 6 | 5
Not completed — Withdrew consent | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Other Miscellaneous Reasons | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LUMIGAN® RC | DuoTrav® | Total
Number analyzed (Participants) | 67 | 68 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (9.7) | 65.2 (10.7) | 66.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: Mean Diurnal Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. The mean diurnal IOP was the average of the IOP values of the study eye (worse eye) at Week 12 measured at 8 AM, 12 Noon and 4 PM. For each study eye, IOP was either the average of 2 measurements, or, if a third measurement was required, the average of 3 measurements.
Time Frame: Week 12
Population: Participants from the modified Intent-to-treat (mITT) population, all randomized participants who received at least one dose of study treatment and met inclusion criteria, with data available for analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LUMIGAN® RC | DuoTrav®
Number analyzed (Participants) | 61 | 63
mmHg | 18.6 (3.5) | 17.4 (2.7)

2. Secondary Outcome: Change From Baseline in Mean IOP at Week 12
Description: IOP is a measurement of the fluid pressure inside the eye. IOP of the study eye (worse eye) was measured at 8 AM, 12 Noon and 4 PM at Week 12. For each eye, IOP was either the average of 2 measurements, or, if a third measurement was required, the average of 3 measurements. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12
Population: Participants from the Full Analysis Set IOP population, all randomized participants who received at least one dose of study treatment and met study inclusion criteria, with IOP data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LUMIGAN® RC | DuoTrav®
Number analyzed (Participants) | 66 | 68
mmHg
  Baseline_8 AM | 22.0 (2.9) | 22.0 (4.1)
  Change from Baseline at Week 12 _8 AM (n=61,63) | -2.7 (3.4) | -4.5 (3.1)
  Baseline_12 Noon | 20.6 (3.2) | 20.3 (3.8)
  Change from Baseline at Week 12_12 Noon (n=61,63) | -1.9 (3.1) | -2.3 (3.2)
  Baseline_4 PM | 19.8 (3.1) | 19.8 (4.1)
  Change from Baseline at Week 12_4 PM (n=61,63) | -1.3 (2.7) | -2.4 (3.5)

3. Secondary Outcome: Percentage of Participants With ≥15% Reduction in Mean Diurnal IOP From Baseline
Description: IOP is a measurement of the fluid pressure in the eye. The mean diurnal IOP was the average of the IOP values of the study eye (worse eye) measured at 8 AM, 12 Noon and 4 PM. For each eye, IOP was either the average of 2 measurements, or, if a third measurement was required, the average of 3 measurements.
Time Frame: Baseline, Week 12
Population: Participants from the mITT population, all randomized participants who received at least one dose of study treatment and met inclusion criteria, with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | LUMIGAN® RC | DuoTrav®
Number analyzed (Participants) | 61 | 63
percentage of participants | 26.2 | 47.6

4. Secondary Outcome: Percentage of Participants With Mean Diurnal IOP Less Than 18 mmHg
Description: IOP is a measure of the fluid pressure in the eye. The mean diurnal IOP was the average of the IOP values of the study eye (worse eye) at Week 12 measured at 8 AM, 12 Noon and 4 PM. For each eye, IOP was either the average of 2 measurements, or, if a third measurement was required, the average of 3 measurements.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | LUMIGAN® RC | DuoTrav®
Number analyzed (Participants) | 61 | 63
percentage of participants | 11.5 | 17.5

5. Secondary Outcome: Change From Baseline in Mean IOP at Week 6
Description: IOP is a measurement of the fluid pressure inside the eye. IOP of the study eye (worse eye) was measured at 8 AM, 12 Noon and 4 PM at Week 6. For each eye, IOP was either the average of 2 measurements, or, if a third measurement was required, the average of 3 measurements. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LUMIGAN® RC | DuoTrav®
Number analyzed (Participants) | 66 | 68
mmHg
  Baseline_ 8 AM | 22.0 (2.9) | 22.0 (4.1)
  Change from Baseline at Week 6 _8 AM (n=66,64) | -2.8 (2.9) | -4.8 (4.1)
  Baseline_12 Noon | 20.6 (3.2) | 20.3 (3.8)
  Change from Baseline at Week 6_12 Noon (n=66,64) | -2.1 (3.1) | -2.8 (3.4)
  Baseline_4 PM | 19.8 (3.1) | 19.8 (4.1)
  Change from Baseline at Week 6_4 PM (n=66,64) | -1.5 (2.5) | -2.9 (3.6)

ADVERSE EVENTS:
Groups:
- Travatan® Z: Travatan® Z (travoprost ophthalmic solution 0.004%) administered as 1 drop in the affected eye(s) once a day for 4 weeks for all participants.
Arm/Group | Travatan® Z | LUMIGAN® RC | DuoTrav®
Serious Adverse Events (participants affected / at risk) | 0/135 | 0/67 | 1/68
Other Adverse Events (participants affected / at risk) | 0/135 | 0/67 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Travatan® Z (N=135) | LUMIGAN® RC (N=67) | DuoTrav® (N=68)
Pyrexia (General disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.